CLINICAL TRIAL: NCT04594902
Title: The PANTHERS (Parents and iNfants Together in Home-based Early Remote Services) Project
Acronym: PANTHERS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: #108696; 1R01HD102201-01 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2020-10-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Early Childhood Development; Behavior Problems
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Randomized control trial in which participants are randomly assigned to either receive the Infant Behavior Program (IBP) or the Enhanced Pediatric Primary Care (EPPC).
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators and coders assessing response over time are kept unaware of the condition to which each participant is assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infant Behavior Program (IBP) (Experimental): Infant Behavior Program (IBP) is a home-based adaptation of the Child-Directed Interaction (CDI) phase of Parent-Child Interaction Therapy (PCIT), an evidence-based intervention for early externalizing problems. Consistent with recommendations we maintained core features of CDI and addressed the unique developmental needs of infants. All IBP sessions will completed remotely.
  Interventions: Behavioral: Infant Behavior Program (IBP)
- Enhanced Pediatric Primary Care (EPPC) (Active Comparator): Families in EPPC will receive six one-hour home visits where they will receive information about normative developmental and health expectations for their infant. Specifically, therapists will provide education on six topics: (1) cognitive and emotional development; (2) language and social development; (3) safety; (4) feeding and nutrition; (5) sleep; and (6) fitness and activity. All EPPC sessions will completed remotely.
  Interventions: Other: Enhanced Pediatric Primary Care (EPPC)

INTERVENTIONS:
Behavioral: Infant Behavior Program (IBP) — Infant Behavior Program (IBP) is a home-based adaptation of the Child-Directed Interaction (CDI) phase of Parent-Child Interaction Therapy (PCIT), an evidence-based intervention for early externalizing problems. Consistent with recommendations we maintained core features of CDI and addressed the unique developmental needs of infants. All IBP sessions will completed remotely.
  Arms: Infant Behavior Program (IBP)
Other: Enhanced Pediatric Primary Care (EPPC) — Families in EPPC will receive six one-hour home visits where they will receive information about normative developmental and health expectations for their infant. Specifically, therapists will provide education on six topics: (1) cognitive and emotional development; (2) language and social development; (3) safety; (4) feeding and nutrition; (5) sleep; and (6) fitness and activity. All EPPC sessions will completed remotely.
  Arms: Enhanced Pediatric Primary Care (EPPC)

SUMMARY:
The PANTHERS (Parents And iNfants Together in Home-based Early Remote Services) Projects is a study funded by the National Institute of Child Health and Human Development to evaluate the efficacy and maintenance of a remote home-based preventive intervention, the Infant Behavior Program (IBP), to decrease behavior problems in infants from high-risk families. All families will participate in five remote evaluations in their home, and families will also receive 6 remote treatment sessions of either the IBP or the EPPC. All participant procedures will be conducted remotely.

DETAILED DESCRIPTION:
Research Design: The proposed study will evaluate the efficacy and maintenance of a remote home-based preventive intervention, the Infant Behavior Program (IBP), to decrease behavior problems in infants from high-risk families. Specifically, the investigators propose to conduct a randomized controlled trial to demonstrate its efficacy and maintenance in reducing behavior problems and increasing infant regulation relative to an enhanced pediatric primary care (EPPC) active control condition. Assessments will occur at pre (week 0)- and post (week 8)-intervention assessments (approximately 2 months apart), as well as at 4-month (week 24) , 8 -month (week 40), and 12-month (week 56) follow-up assessments.

Procedures: Families will be primarily recruited from pediatric primary care centers and will be randomized to receive six sessions of either IBP or EPPC in their home. Families also will participate in five remote home-based assessments.

Risks and Benefits: Families may experience risk from a breach in confidentiality as participants reveal sensitive information and there are risks in breach of confidentiality due to videoconferencing methods, in particular if study staff become aware of abuse or neglect situations. Families may experience discomfort when answering personal questions. Benefits to families could include providing families with information that can assist in caring for their child, and instilling new parenting strategies that are designed to outlast treatment.

Knowledge: This study will provide information about the efficacy of a remote home-based preventive intervention to improve infant behavior and regulation.

ELIGIBILITY:
Inclusion Criteria:

* Infants ages 12 to 18 months and at least one primary caretaker, who is at least 18-years-old and in most cases will be the mother
* Elevated score (> 75th percentile) on the problem scale of the Brief Infant-Toddler Social and Emotional Assessment (BITSEA; Briggs-Gowan et al., 2004)
* An English-speaking or Spanish-speaking primary caregiver.

Exclusion Criteria:

* Infants with major sensory impairment (e.g., deafness blindness) or several problems that impair mobility (e.g., cerebral palsy)
* Significant cognitive delay in the primary caregiver (i.e., estimated IQ score < 70 on the vocabulary subtest of the Wechsler Abbreviated Scale of Intelligence - Second Edition (WASI-II) for those speaking English or an average standard score < 4 on the vocabulary subtest of the Escala de Inteligencia Wechsler Para Adultos - Third Edition (EIWA-III) for those speaking Spanish)
* Families involved with child protection services, which is expected to be low based on our pilot trials

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 288 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-09-07 (Estimated); Study Completion 2026-09-07 (Estimated)

PRIMARY OUTCOMES:
Infant-Toddler Social and Emotional Assessment (ITSEA) | Change from week 0 to weeks 8, 24, 40, and 56
  The ITSEA is a 166-item parent-report measure of the frequency of specific behaviors (e.g., temper tantrums) in 12- to 36-month-olds. Participants will score their child behavior on a scale of 0-2 (0 Not true/Rarely, 2 Somewhat True/Sometimes and 3 Very True/Often). The higher the score, the higher the child is on behavior problems. The Externalizing scale will be an indicator of infant behavior. The higher the score the higher child's behavior problems.

SECONDARY OUTCOMES:
Wechsler Abbreviated Scale of Intelligence Second Edition (WASI-II) | Screen
  The WASI will be used at screening to ensure ability to learn the skills. The vocabulary and matrix reasoning subtests will be administered, and primary caregivers will be required to receive an estimated IQ score ≥ 70 on the two-subtest version of the WASI-II. The higher the score the higher IQ.
Brief Infant-Toddler Social Emotional Assessment (BITSEA) | Screen
  The BITSEA will be used at screening as inclusion criteria. The 31-item Problem scale will be used to screen infants for the inclusion criterion (≥ 75th percentile) because it has high sensitivity and specificity in detecting current and predicting subsequent elevated externalizing problems. The higher the score the higher the child's behavior problem.
Ages and Stages Questionnaire-Third Edition (ASQ-III) | Week 0
  Assess for developmental delay in children ages three months to five years. It is a 30-item parent-rating scale used to assess for developmental delay in children ages three months to five years. The ASQ-III has high test-retest reliability, interrater reliability, and concurrent validity134 and will be used as a baseline measure of the infant's developmental functioning. We will administer every scale- communication, gross motor, fine motor, problem solving, personal-social. Families respond to various milestones prompts on a scale of Yes, Sometimes, Not Yet. The higher the score the the higher the outcome.
Dyadic Parent-Child Interaction Coding System-IV (DPICS-4) | Change from weeks 0 to week 8, 24, 40, and 56
  The Dyadic Parent-Child Interaction Coding System-4th Ed (DPICS-IV; Eyberg et al., 2013) is a structured behavioral observation coding system assessing caregiver-child interactions. Observed parenting behaviors will be coded during a 5-min child-led play and combined into two categories of positive (praises, behavior descriptions, and reflections) and negative (questions, commands, and negative talk) verbalizations, reflecting behaviors caregivers are taught to use and avoid in PCIT. Additionally, child compliance will be assessed and coded for during a 5-min caregiver-led play and 5-min clean up situation which will be adapted to meet the infant's developmental level (e.g., toy bucket in close proximity to infant). The higher the score the higher the parenting behavior and child compliance.
Early Childhood Behavior Questionnaire-Very Short Form (ECBQ) | Change from weeks 0 to week 8, 24, 40, and 56
  The ECBQ is a 36-item parent questionnaire of temperament. The effortful control scale will be used as the behavioral indicator of infant regulation. Participants will respond to various child behavior prompts using the 1-7 scale: 1- never, 2-very rarely, 3- less than half the time, 4- about half the time, 5- more than half the time, 6- almost always, 7- always. The higher the score the higher the outcome.
Laboratory Temperament Assessment Battery (Lab-TAB) | Change from weeks 0 to week 8, 24, 40, and 56
  The Lab-TAB is a standardized observation to assess early regulation. We will include an episode to elicit mild frustration that will involve the infant playing with a desired toy for 30 seconds, and then the parent will remove the toy from the infant and place the toy in a clear box that the child cannot open for 1 minute (repeated twice). Episodes will be videotaped and coded for infant emotional reactivity (latency to distress in seconds), lability (range from 0 = unstable to 4 = stable), and regulation (range from 0 = dysregulated to 4 = well-regulated). The higher the child distress the higher the outcome.
Short-form version of the MacArthur Communicative Development Inventories | Change from weeks 0 to week 8, 24, 40, and 56
  The MacArthur Short-form is an 89-word checklist for infant vocabulary comprehension and production and completed by the primary caregiver. Participants indicate which of a prespecified list of words the child can already understand and/or produce. The full scale will be administered, and the higher the score the higher the child's vocabulary.
Brief Infant Sleep Questionnaire (BISQ) | Change from weeks 0 to week 8, 24, 40, and 56
  10-item questionnaires used to measure infant and toddler sleep problems. There are no scales in this questionnaire.
Screen Media Use Questionnaire A | Week 0
  The Screen Media Use Questionnaire A is a 6 item questionnaire to obtain information on family usage of screen devices. There are no scales in this questionnaire.
Screen Media Use Questionnaire B | Repeated at weeks 8, 24, 40, and 56.
  The Screen Media Use Questionnaire B is a 21 item questionnaire to obtain information on family usage of screen devices. There are no scales in this questionnaire.
Screen Media Use Interview | Repeated at weeks 0, 8, 24, 40, and 56.
  The Screen Media Use Interview was development by our team to obtain information of caregiver and infant use of screens (e.g., amount of time on screens, type of screen use). There are no scaled in this questionnaire.
Parenting Scale | Change from weeks 0 to week 8, 24, 40, and 56
  The Parenting Scale is a 30-item self-report of parenting practices. Participants report their parenting strategies by answering prompts on 7-point likert scales. 1 indicates a high probability of using an effective discipline strategy and 7 indicates a high probability of ineffective discipline The Overreactivity scale will be used as an indicator of negative parenting practices. The higher the score the higher the outcome.
Parental Sensitivity/Responsivity: Global codes from the Early Parenting Coding System (EPCS) | Change from weeks 0 to week 8, 24, 40, and 56
  Global codes from the Early Parenting Coding System (EPCS), will be used to rate parental sensitivity/responsivity during the five-minute play. This is an observational tool with no scales.
Positive and Negative Affective Schedule (PANAS) | Change from weeks 0 to week 8, 24, 40, and 56
  The Positive and Negative Affective Schedule (PANAS) is a 20-item self-report measure (10 positive and 10 negative affective descriptors) with strong psychometric properties.The negative affect scale measures emotional experiences common to depression and anxiety and will be used as an indicator of parental distress. Participants respond with a 1-5 scale: 1- very slightly or not at all, 2- a little, 3- moderately, 4- quite a bit, 5- extremely. The higher the score the higher the outcome.
The Parenting Stress Index, Fourth Edition Short Form (PSI-SF) | Change from weeks 0 to week 8, 24, 40, and 56
  The PSI-SF parental distress scale will be used as an indicator of parental distress. The PSI-SF is a 36-item self-report questionnaire of parenting stress with three subscales (PD, PCDI, and DC) and a Total Stress scale. Families rate the responses with a likert-like scale: SA- Strongly Agree, A- Agree, NS- Not Sure, D- Disagree, SD- Strongly Disagree. The higher the score the higher the outcome.
Abbreviated Multidimensional Acculturation Scale (AMAS) | Week 0
  The AMAS will be used to assess acculturation. It is a 42-item scale with 4-point self-report, Likert-type response options ranging from 1(strongly disagree) to 4 (strongly agree) for the cultural identity subscales and from 1 (not at all) to 4 (extremely well/like a native) for the language and cultural competence subscale. High scores relate to higher the acculturation..
Multidimensional Acculturative Stress Inventory (MASI) | Week 0
  The MASI will be used to assess acculturative stress. Families rate their responses to prompts across four scales (Spanish Competency Pressures, English Competency Pressures, Pressure to Acculturate and Pressure Against Acculturation) on a 0-5 likert scale (0- Not Applicable, 1- Not at all stressful, 2- A little stressful, 3- Somewhat stressful, 4- Very stressful, 5- Extremely stressful). All the scales will be administered, and the higher the score the higher the outcome.
Adult Executive Functioning Inventory (ADEXI) | Week 0
  The ADEXI requires that the informant rate the extent to which each item is true about them on a 5-point Likert scale (1: Definitely not true, 5: Definitely true). The questions are related to the frequency with which the informant experiences difficulty related to working memory and inhibition in everyday life. The higher the score the higher the outcome.
NIH Cognitive Toolbox List Sorting Working Memory Test | Week 0
  The List Sorting Working Memory Test assesses ability to store information until the amount of information to be stored exceeds one's capacity to hold that information. This is an observational task.
Services for Children and Adolescents-Parent Interview (SCAPI) | Change from weeks 0 to week 8, 24, 40, and 56
  The SCAPI is a structured parent interview providing information on the type, number, duration, and intensity of physical and mental health services provided for the child and will be used to control for group differences in additional services families received in between each assessment, if applicable. The interview asks if the child has received any of the following services: Speech/Language Therapy, Physical Therapy, Occupational Therapy, Sensory Integration Therapy, Individual Child Counseling for Behavioral or Emotional Problems, Parent Training, Family Therapy, Play Therapy, Group Counseling. There are no scaled responses.
Technological Ease and Computer-based Habits Inventory (TECHI) | Week 0
  The TECHI assesses caregiver and child technology use and literacy as a potential moderator of treatment response. Participants rate their comfort level with technology on a Strongly Disagree- Strongly Agree 0-5 likert scale. The higher the score the higher the comfort level with technology. The entire inventory will be administered.
Therapy Attitude Inventory (TAI) | Week 8
  The TAI is used document satisfaction with the intervention. The higher the score the higher the therapy satisfaction.
IBP Quiz | Week 8
  The IBP quiz will be administered to the IBP group only. The quiz was developed to asses parent's understanding of the information received during their participation in the program. The higher the score the higher the understanding.
EPPC Quiz | Week 8
  The EPPC quiz will be administered to the EPPC group only. The quiz was developed to asses parent's understanding of the information received during their participation in the program. The higher the score the higher the understanding.
Center for Epidemiologic Studies Depression Scale (CES-D) | Change from weeks 0 to week 8, 24, 40, and 56
  The Center for Epidemiologic Studies Depression Scale (CES-D) is a 20-item self-report measure of depressive symptoms with strong psychometric support. The CES-D total score will be used as an indicator of parental distress. Participants respond to predetermined statements on a Likert-like scale. The higher the score the higher the depression symptoms.
COPING WITH TODDLERS' NEGATIVE EMOTION SCALE (CTNES) | Change from weeks 0 to week 8, 24, 40, and 56
  The Coping with Toddlers' Negative Emotions Scale (CTNES)161 is a measure of parent response to child negative emotions with support for use with infants.162 Consistent with previous work,163 we will combine items on the problem-focused, emotion-focused, and expressive-encouragement subscales as an indicator of parental responsivity. The higher the score the higher the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Bagner, PhD, Principal Investigator — Florida International University
Locations (2):
- United States (2):
  - South Miami Children's Clinic, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
We will use a controlled access approach, using a robust system to review requests and provide secure access to de-identified data
Supporting Information: Study Protocol
Time Frame: Deidentified data for the entire database will be made available for data sharing after the main findings from the final dataset have been accepted for publication.
Access Criteria: Users will be provided with the data under a data-sharing agreement which specifies that: (1) data will be used only for research purposes; (2) data will be stored confidentially and securely; and (3) data will be destroyed after analyses are completed. PI Bagner and collaborators will identify where the data will be available and how to access the data in any publications and presentations using these data.

REFERENCES:
- [Background] Bagner DM, Coxe S, Hungerford GM, Garcia D, Barroso NE, Hernandez J, Rosa-Olivares J. Behavioral Parent Training in Infancy: A Window of Opportunity for High-Risk Families. J Abnorm Child Psychol. 2016 Jul;44(5):901-12. doi: 10.1007/s10802-015-0089-5. PMID 26446726
- [Background] Heymann P, Heflin BH, Baralt M, Bagner DM. Infant-directed language following a brief behavioral parenting intervention: The importance of language quality. Infant Behav Dev. 2020 Feb;58:101419. doi: 10.1016/j.infbeh.2019.101419. Epub 2020 Jan 9. PMID 31927404
- [Background] Garcia D, Rodriquez GM, Hill RM, Lorenzo NE, Bagner DM. Infant Language Production and Parenting Skills: A Randomized Controlled Trial. Behav Ther. 2019 May;50(3):544-557. doi: 10.1016/j.beth.2018.09.003. Epub 2018 Sep 11. PMID 31030872
- [Background] Morningstar M, Garcia D, Dirks MA, Bagner DM. Changes in parental prosody mediate effect of parent-training intervention on infant language production. J Consult Clin Psychol. 2019 Mar;87(3):313-318. doi: 10.1037/ccp0000375. Epub 2018 Dec 27. PMID 30589352
- [Background] Blizzard AM, Barroso NE, Ramos FG, Graziano PA, Bagner DM. Behavioral Parent Training in Infancy: What About the Parent-Infant Relationship? J Clin Child Adolesc Psychol. 2018;47(sup1):S341-S353. doi: 10.1080/15374416.2017.1310045. Epub 2017 Apr 17. PMID 28414546
- [Background] Ramos G, Blizzard AM, Barroso NE, Bagner DM. Parent Training and Skill Acquisition and Utilization Among Spanish- and English-Speaking Latino Families. J Child Fam Stud. 2018 Jan;27(1):268-279. doi: 10.1007/s10826-017-0881-7. Epub 2017 Oct 17. PMID 29456439
- [Background] Bagner DM, Garcia D, Hill R. Direct and Indirect Effects of Behavioral Parent Training on Infant Language Production. Behav Ther. 2016 Mar;47(2):184-97. doi: 10.1016/j.beth.2015.11.001. Epub 2015 Nov 14. PMID 26956651
- [Background] Bagner DM, Rodriguez GM, Blake CA, Rosa-Olivares J. Home-Based Preventive Parenting Intervention for at-Risk Infants and Their Families: An Open Trial. Cogn Behav Pract. 2013 Aug 1;20(3):334-348. doi: 10.1016/j.cbpra.2012.08.001. PMID 25414568